CLINICAL TRIAL: NCT05191901
Title: The EFFECT of STRESS BALL on REDUCING the FEAR and PAIN OCCURRENT DURING the PROCEDURE in CHILDREN
Brief Title: The EFFECT of STRESS BALL DURING the PROCEDURE in CHILDREN
Acronym: Stress ball
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ayse Sonay Turkmen, Prof.Dr (Other)
Responsible Party: Sponsor-Investigator, Ayse Sonay Turkmen, Prof.Dr, Assoc.Prof., Karamanoğlu Mehmetbey University
Organization: Karamanoğlu Mehmetbey University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Stress Ball
Record Dates: First submitted 2021-12-20; First posted 2022-01-14 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2022-05

CONDITIONS: Having a Blood Draw
Keywords: Pain; Turning Attention; Establishing intravascular access; Fear
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- stress ball group (Experimental)
  Interventions: Other: Stress Ball
- control group (No Intervention)

INTERVENTIONS:
Other: Stress Ball — Reducing pain and fear by squeezing a stress ball during the blood draw procedure.
  Arms: stress ball group

SUMMARY:
This research was planned in a Randomized Controlled Experimental Research design with Pre-Test-Post-Test Control Group in order to determine the effect of the stress ball squeezing technique applied to children aged 7-12 during the vascular access procedure on the level of fear and pain in children. The data of the study were obtained from children aged 7-12 who came to the Karaman Training and Research Hospital Pediatrics Service between August 1 and October 31, 2020. The sample size was determined as 116 children in total, 58 children for each group. "Interview and Observation Form, Children's Fear Scale (CFS), Wong-Baker Faces, Stress Ball and Stopwatch" were used for data collection.

In order to evaluate whether the research is ethically appropriate, an application was made to the Ethics Committee of Karamanoğlu Mehmetbey University School of Health Sciences and the necessary permission was obtained. Written permission was obtained from the Chief Physician of Karaman Training and Research Hospital in order to conduct the study in the Child Health and Diseases Service of Karaman Training and Research Hospital.

Statistical analyzes of the study will be done in SPSS 21.0 package program. Number, percentage, mean and standard deviation values will be used from descriptive analyses. In the analysis of differences between groups, independent groups t test, paired t test, Anova, Mann Whitney U and Kruskal Wallis tests will be used. Tukey or Duncon tests will be used for further analysis. The change in the post-procedural pain level of children according to some variables will be evaluated with multiple and simple regression analyses. Significance level will be accepted as p<0.05.

DETAILED DESCRIPTION:
Dependent variable: Children's level of pain and fear Independent variable: Stress ball, demographics, previous painful transaction experience Randomization of control and stress ball groups; The status of the children to be included in the study in the control or stress ball group was determined by using "stratification and randomization methods with blocks". In the literature, it has been reported that gender and fear of interventional procedures are among the factors affecting the fear and anxiety experienced by children in interventional procedures (Törüner & Büyükgönenç, 2012; Çavuşoğlu, 2013). Accordingly, stratified and block randomization will be applied to the children as "girl and boy" for the gender variable and "afraid and not afraid" for the fear of the procedure. 58 children will be included in each of the research groups. During the data collection process, each child and family will be taken to the invasive procedure room individually. This will prevent children from meeting with each other.

The determined layers were created by the statistician as codes obtained from a permutation-based computer program (https://www.randomizer.org). At the beginning of the study, which letter would be the stress ball or the control group was determined by the closed opaque envelope method, and the letter A was used for the stress ball group and the letter B was used for the control group.

Blinding: Single blinding (participants) will be used in the study. Participants will not be told whether they are in a stress ball or control group. A separate informed consent form will be created and approved for each group. In order to prevent children and parents from encountering each other, information will be given in the closed operation room and their consent will be obtained. Each child will be taken to a separate room with one of their parents. It will be ensured that no child is waiting near the door for invasive intervention.

Hypotheses H0: The stress ball applied during the vascular access procedure does not affect the fear and pain levels of children.

H1: The stress ball applied during the venipuncture procedure affects the children's fear levels H2: The stress ball applied during the vascular access procedure affects the pain levels of children.

H3: The stress ball applied during the venipuncture procedure affects the satisfaction of children, parents and nurses.

The research will be carried out in the following order.

1. Since the vascular access procedure will be performed by a single nurse, the children who are admitted to the service during the working day and time of the determined nurse and those whose parents are volunteers will be included in the study. Before the data collection phase, children and parents who meet the sample selection criteria of the research will be informed about the purpose and content of the research, and verbal and written consent will be obtained from their parents.
2. Materials will be prepared beforehand (data collection tools, stress ball, stopwatch).
3. Individual characteristics will be obtained from children and family members and recorded in the interview and observation form. Before the procedure, the fear level of children about the procedure will be recorded by asking the child, parent and observer separately using the Children's Fear Scale (CFS).
4. The status of the child in the stress ball or control group will be determined by using layer sets.
5. Children in the control group will be taken to the invasive procedure room and a parent will be with the child during the vascular access procedure. During the procedure, as soon as the children start to cry, the stopwatch will be started and will continue to run throughout the crying. After the procedure, the child's fear (Children's Fear Scale (CFS)) and pain (Wong-Baker FACES) related to the procedure will be evaluated separately by the child, parent and observer and recorded in the form.
6. Children in the stress ball group will be asked to hold and squeeze the stress ball in their untreated hands before starting the vascular access process. A parent will be provided with the child during the procedure. A few seconds after the child starts squeezing the ball, the vascular access process will be started. The child will be asked to continue the process of squeezing the ball until the intravenous access is completed. During the procedure, as soon as the children begin to cry, the stopwatch will be started and will continue to run throughout the crying. After the procedure, the child's fear (Children's Fear Scale (CFS)) and pain (Wong-Baker FACES) related to the procedure will be evaluated separately by the child, parent and observer and recorded in the form.

ELIGIBILITY:
Inclusion Criteria:

* The child is between the ages of 7-12
* Absence of pain (due to disease, drug side effects, distension)
* Absence of any physical or mental illness
* Being able to communicate and being open to communication
* No history of ischemic epilepsy, migraine or vestibular disorder
* No long-term illness.
* Absence of a regularly used medication
* Not taking analgesics in the last six hours
* Hospitalization for diagnosis or treatment
* Vascular access is performed by the same nurse,
* Single way vascular access
* The child and parent speak and understand Turkish comfortably,
* The child and his parents do not accept to participate in the study, and they do not have a speech or vision disorder.

Exclusion Criteria:

* who do not meet the inclusion criteria.

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 116 (Actual)
Dates: Start 2022-03-14 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-05-20 (Actual)

PRIMARY OUTCOMES:
Pain scores | 5 minutes
Fear scores | 5 minutes

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - KaramanogluMehmetbeyU, Karaman, Turkey
  - Karamanoglu Mehmetbey University, Karaman

IPD SHARING:
Plan to Share IPD: No